CLINICAL TRIAL: NCT06637475
Title: Investigation of the Effects of External Electrical Stimulation in Women With Vaginal Laxity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Zehra KORKUT, Asst. Prof., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZKORKUT
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Vaginal Laxity
Keywords: vaginal laxity, pelvic floor, electrical stimulation
MeSH Terms: interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: Individuals who meet the inclusion criteria and who have signed the consent form will be randomly divided into 2 groups (treatment and control groups). Randomization will be done by a researcher who is not involved in the study using computer-assisted randomization blocks. The treatment group patients will receive 3 sessions of external stimulation per week for 8 weeks, while the control group will not receive any intervention (consisting of patients waiting on the treatment list).
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- electric stimulation group (Experimental): Individuals who meet the inclusion criteria and who have signed the consent form will be randomly divided into 2 groups (treatment and control groups). Randomization will be done by a researcher who is not involved in the study using computer-assisted randomization blocks. The treatment group patients will receive 3 sessions of external stimulation per week for 8 weeks, while the control group will not receive any intervention (consisting of patients waiting on the treatment list).
  Interventions: Device: Electric stimulation
- control group (No Intervention)

INTERVENTIONS:
Device: Electric stimulation — Patients with baseline assessments will be followed up for 8 weeks within a planned treatment program. Treatment protocol for the ES group:
  external ES wearable apparatus will be applied three days a week for 30 minutes with symmetrical biphasic current at a frequency of 50 Hertz (Hz), with stimulation and rest periods of 5 s contraction and 5 s rest, with a current intensity ranging from 0-100 mA while the patients are in the supine position. The device will be attached to the patients in such a way that it wraps around the upper thigh, the electrodes will be attached to the anterior and posterior of the right and left thigh, the right-left pelvic side and the right-left gluteal region. The current intensity in each session will be determined as the maximum current intensity that will not cause pain and discomfort in individuals.
  Arms: electric stimulation group

SUMMARY:
The aim of this study was to investigate the effects of external electrical stimulation on clinical symptoms such as vaginal symptoms, pelvic floor symptoms, sexual function, pelvic floor muscle morphometry (levator ani thickness) and functions (strength, endurance), vaginal wall thickness and perception of healing in women with vaginal laxity.

ELIGIBILITY:
Inclusion Criteria:Complaining of vaginal laxity To be between 18-60 years old, Being sexually active, Volunteering to participate in the study, Becoming literate -

Exclusion Criteria:

Sensory loss Presence of infection Having a pacemaker Metal implant presence Malignancy story Having serious cardiovascular problems Presence of severe pelvic organ prolapse (above stage 2) Having undergone surgery for POP/incontinence (within the last 1 year) Pregnancy presence Having enough laxity to require surgery Having a neurological disorder Receiving estrogen therapy

-

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Vaginal Symptoms International Consultation on Incontinence Questionnaire - Vaginal Symptoms (ICIQ-VS) | Change from basline at 8 weeks

SECONDARY OUTCOMES:
Pelvic floor symptoms Pelvic Floor Distress Inventory-20 (PTDE-20) | Change from basline at 8 weeks
Sexual function Female Sexual Function Index (FSFI) | Change from baseline at 8 weeks
Pelvic floor muscle morphometry (levator ani thickness) | Change from baseline at 8 weeks
Pelvic floor muscle strength and endurance | Change from baseline at 8 weeks
Vaginal wall and mucosa thickness | Change from basline at 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No